CLINICAL TRIAL: NCT01196247
Title: Stand Up to Cancer Consortium: Phase II Study of Therapy Selected by Molecular/Metabolic Profiling in Patients With Previously Treated With Metastatic Pancreatic Cancer
Brief Title: A Study of Therapy Selected by Molecular/Metabolic Profiling in Patients With Previously Treated Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Drug Development (Other)
Collaborators: Scottsdale Healthcare (Other); Stand Up To Cancer (Other); American Association for Cancer Research (Other)
Responsible Party: Ramesh Ramanathan, MD, TGen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU2C-001
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Previously Treated Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; molecular profiling; SU2C; Second line therapy; Stage 4
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Comparative Genomic Hybridization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Drug will be recommended based on IHC/Fish, CGH and Pan-XenoBank — FDA approved drugs as indicated by molecular profiling
  Other Names: FDA approved drugs as indicated by molecular profiling

SUMMARY:
The purpose of the study is selecting second line therapy for patients with pancreatic cancer using molecular profiling will improve 1 year survival.

DETAILED DESCRIPTION:
Following first-line therapy with a gemcitabine based regimen, a significant number of patients will maintain an adequate performance status and be able to tolerate a second-line therapy. A recent phase III trial randomized patients to either 5-flurouracil (5FU), folinic acid or to the addition of weekly oxaliplatin to the same regimen of 5FU/folinic acid. The interim results showed a statistically significant survival advantage for the oxaliplatin containing arm (26 versus 13 weeks, P= 0.014). However the outcome of patients who have progressed on a first-line gemcitabine regimen is still poor with median survival of about 2-6 months.

Almost all patients with advanced APC, treated with gemcitabine alone or a gemcitabine based combination therapy will exhibit resistance to therapy. In patients treated with gemcitabine alone, the time to progression (TTP) is about 3-4 months. Thus most patients will exhibit progression and /or toxicity and will require second line therapy at 4-6 months into first line therapy. The best one year survival reported in a phase II trial is only 24%. However there is no standard second line therapy for APC, a rapid progression of tumor is seen in this setting, and new strategies based on rational target identification are needed. In this study we propose to select therapy based on the molecular profiling of each patients tumor.

ELIGIBILITY:
Inclusion Criteria:

* metastatic adenocarcinoma of the pancreas
* male or non-pregnant female
* 18 years of age or greater
* one prior therapy for the treatment of metastatic disease
* must start continuation therapy within 9 months of starting first line treatment
* have adequate organ and bone marrow function
* must have a Karnofsky performance status greater than or equal to 70
* one or more metastatic tumors measurable by CT scan and accessible for biopsy

Exclusion Criteria:

* operable or locally advanced pancreatic cancer
* metastatic tumor that is not amendable to biopsy
* known brain mets unless previously treated and well controlled
* active, uncontrolled bacterial, viral or fungal infections
* known infection with HIV, hepatitis B or hepatitis C
* pregnant or breast-feeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Determine the percent of patients who are alive at one year | One year
  Goal is to improve the one year survival (from start of first-line therapy for metastatic disease) to 60%

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, MD, Principal Investigator — TGen
Locations (1):
- TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona, United States